CLINICAL TRIAL: NCT01814085
Title: A Single-arm, Open-label, Multi-center Study to Investigate Efficacy and Safety of Lexapro on Acute Treatment of Severe Depression
Brief Title: A Safety and Efficacy Study of Escitalopram on Acute Treatment of Severe Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016300; ESCITALDEP4001
Record Dates: First submitted 2013-03-14; First posted 2013-03-19 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Escitalopram; Lexapro
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Experimental): Escitalopram tablets will be administered orally in the dose range of 10 to 20 milligram per day (mg/day) for 8 weeks. Dose can be adjusted as per Investigator's discretion depending on participant's response.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram tablets will be administered orally in the dose range of 10 to 20 milligram per day (mg/day) for 8 weeks. Dose can be adjusted as per Investigator's discretion depending on participant's response.
  Other Names: Lexapro

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of escitalopram treatment in participants with severe major depressive disorder (MDD [marked depression appearing in the involution period and characterized by hallucinations, delusions, paranoia, and agitation]).

DETAILED DESCRIPTION:
This is a single-arm (clinical study in only one group of participants), open-label (all people know the identity of the intervention), multi-center (when more than one hospital or medical school team work on a medical research study), and prospective (study following participants forward in time) study. The study consists of 2 parts: Screening (that is, 5 days before study commences on Day 1) and Treatment (that is, Week 1-8). All the eligible participants will be receiving flexible doses of escitalopram orally in the dose range of 10 to 20 milligram per day (mg/day) for 8 weeks. Efficacy will primarily be evaluated by remission rate at the end of the study. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with major depressive disorder (MDD) according to Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV)
* Scores of greater than or equal to 30 on the Montgomery-Asberg Depression Rating Scale (MADRS) Exclusion Criteria:
* Pregnant or lactating female participants
* Participants who are previously or currently diagnosed with the following mental disorders by DSM-IV: organic mental disorder, schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self), schizoaffective disorder, delusional disorder, undifferentiated mental disorders and bipolar affective disorder, participants with history of drug abuse, including alcohol and drug abuse in the past 12 months
* Participants who have significant risk of suicide on clinical assessment (has a score of greater than or equal to 5 on item 5 of MADRS) or have made a serious suicide attempt within the past 6 months and have any contraindication to escitalopram
* Participants who have known history of serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease currently taking other psychotropic drugs and anticonvulsant agents or continuously taking benzodiazepines or sleeping pills for over five days in the past one week
* Participants who have history of seizure (sudden, uncontrolled muscle spasms and loss of consciousness resulting from abnormal brain function) disorder, brain injury, any history of known neurological disease (multiple sclerosis, degenerative diseases, parkinson disease and any movement disorders) and have multiple drug adverse reactions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Remission Based on Montgomery-Asberg Depression Rating Scale (MADRS) | Week 8
  Remission is defined as percentage of participants with MADRS total score less than or equal to10 at the endpoint (8 weeks). The MADRS is a scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher score represents a more severe condition.

SECONDARY OUTCOMES:
Percentage of Participants With Clinical Response Based on Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline and Week 8
  Clinical response is defined as greater than or equal to 50 percent change from Baseline in MARDS total scores at end point (8 weeks). The MADRS is a scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher score represents a more severe condition.
Percentage of Participants With Clinical Onset Based on Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline and Week 8
  Clinical onset is defined as the reduction rate of MADRS total score greater than or equal to 20 percent. The MADRS is a scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher score represents a more severe condition.
Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 1, 2, 4 and 8 | Baseline, Week 1, 2, 4 and 8
  The MADRS is a scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher score represents a more severe condition.
Change From Baseline in Hamilton Depression Rating Scale (HAM-D-17) Score at Week 1, 2, 4 and 8 | Baseline, Week 1, 2, 4 and 8
  The Hamilton Depression Rating (HAM-D-17) Scale is a 17-item scale used to assess the severity of depression in participants diagnosed with an affective disorder. Items are scored from 0 to 4, the higher the score, the more severe the depression. Questions are related to symptoms such as depressed mood, guilt feelings, suicide, sleep disturbances, anxiety levels and weight loss.
Change From Baseline in Hamilton Anxiety Scale (HAMA) Score at Week 1, 2, 4 and 8 | Baseline, Week 1, 2, 4 and 8
  The Hamilton Anxiety Rating (HAMA) Scale is a 14-item scale developed to measure the severity of symptoms such as anxiety, tension, depressed mood, palpitations, breathing difficulties, sleep disturbances, restlessness and other physical symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe).
Change From Baseline in Brain-Derived Neurotrophic Factor (BDNF) at Week 8 | Baseline and Week 8
  Serum BDNF levels normally decrease in participants suffering from Major Depressive Disorder (MDD) and the decrease is more prominent in participants with long disease course but this can also increase in response to antidepressants. The enzyme-linked immunosorbent assay (ELISA) method will be used to evaluate the serum BDNF level before and after using escitalopram, and use it as a biological marker for predicting the early efficacy of taking antidepressants.
Change From Baseline in Short Form-12 (SF-12) Score at Week 8 | Baseline and Week 8
  The SF-12 health survey is the 12-item sub form of Short form (SF-36), investigating 8 health dimensions: physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. This 12-item scale measures health conditions and describes the level of general physical health state and mental health problems.
Change from Baseline in Plasma Drug Concentration at Week 1 and 8 | Baseline, Week 1 and 8
  Plasma concentration of study drug will be assessed in blood samples.
Number of Participants with Structural and Functional Changes in Magnetic Resonance Imaging (MRI) at Week 8 | Baseline and Week 8
  Major depressive disorder participants have distinctive prefrontal cortex, hippocampal atrophy (wasting away, or decrease in size, of a body organ) and amygdala function abnormalities. Structural and functional MRI (body pictures created using magnetic waves to look at soft tissues of the body) can help to evaluate the efficacy of escitalopram on neural plasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (6):
- China (6):
  - Beijing
  - Huzhou
  - Nanjing
  - Qingdao
  - Shanghai
  - Wuhan

REFERENCES:
- See also: A Single-arm, Open-label, Multi-center Study to Investigate Efficacy and Safety of Lexapro on Acute Treatment of Severe Depression — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2340&filename=CR016300_CSR.pdf